CLINICAL TRIAL: NCT06705855
Title: A Comparison of Renal vs Limb NIRS for Predicting Cardiac Surgery Associated Acute Kidney Injury
Status: Recruiting | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Natalie Silverton, Associate Professor of Anesthesiology, University of Utah
Other Study IDs: 00179157
Record Dates: First submitted 2024-11-19; First posted 2024-11-26 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: NIRS; Cardiac Surgery Associated - Acute Kidney Injury; Cardiac Surgery Requiring Cardiopulmonary Bypass; AKI - Acute Kidney Injury
Keywords: Cardiovascular
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Adult cardiac surgery patients undergoing cardiopulmonary bypass surgery at risk for AKI: We will enroll a convenience sample of adult cardiac surgery patients undergoing procedures that require cardiopulmonary bypass (CPB) and who are at risk for AKI.
  Interventions: Device: NIRS sensor placement

INTERVENTIONS:
Device: NIRS sensor placement — After written informed consent, the patient will be brought to the operating room. Skin tone will be assessed using the Monk scale. Prior to induction of general anesthesia, the right kidney will be located by surface ultrasound, the distance between the renal capsule and the skin will be measured, and a NIRS sensor will be placed on the skin overlaying the kidney. If the patient has had a right nephrectomy, the left kidney will be used. Additional NIRS sensors will then be placed over the patient's ipsilateral biceps and vastus lateralis muscles. The distance from the skin to the muscle tissue will be measured and recorded using ultrasound. NIRS sensors will also be placed on the patient's forehead to measure cerebral oximetry as is current practice at our institution for all cardiac surgeries requiring cardiopulmonary bypass.

SUMMARY:
Acute kidney injury (AKI) is a complication of cardiac surgery that can affect outcome. Near Infrared Spectroscopy (NIRS) is a technology that uses light to determine how well oxygenated tissues are. This technology is routinely used in cardiac surgery to measure the oxygen level in the brain by placing a sensor sticker on the forehead. The purpose of the study is to determine whether NIRS sensor stickers placed on the skin over the kidney can predict AKI better than when sensors are placed on the skin over the participant's limbs. This study is being conducted by investigators from the department of anesthesiology at the University of Utah.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common complication of cardiac surgery occurring in up to 40% of patients.1, 2 This is more than 10 times the rate of other serious post-surgical complications in cardiac surgery such as stroke or deep sternal infection and is even greater than the incidence of prolonged ventilation.3, 4 Severe AKI requiring new onset dialysis after cardiac surgery occurs in 1-6% of cardiac surgery patients.3, 5 AKI increases length of hospital stay from 5 to 11 days and increases hospital costs from $18,463 to $37,674 per patient.6 The severity of AKI is strongly associated with in-hospital mortality with even the mildest forms of AKI having more than double the mortality and the more severe forms having 10-30 times higher mortality rates (depending on the definition of severe AKI and the patient population).6, 7 AKI contributes to 300,000 annual deaths in the U.S. and 2 million deaths globally each year.8, 9 Considering only the most relevant patient populations (major aortic and spinal surgery, relevant cardiovascular procedures, intensive care patients on mechanical ventilation, severe trauma patients), in the US alone more than 3.1 million patients per year are at risk of AKI.10-14 Of those, 30.6%12, 13, 15 will suffer AKI - adding annual hospital costs of $19 billion.6 It is for these reasons that the Society of Thoracic Surgeons lists renal failure as one of the 5 major complications of cardiac surgery.

The pathophysiology of AKI after cardiac surgery is multifactorial but the profound hemodynamic changes that occur in cardiac surgery likely play an important role. The renal medulla has the highest metabolic activity and least oxygen reserve in the kidney and medullary hypoxia is thought to be a major determinant of AKI.16, 17 One major limitation in the effort to reduce the incidence of AKI is the lack of a real-time monitor of renal hypoxia. As there is no current therapy for AKI once the disease has occurred, prevention is the mainstay of treatment and an important step in preventing AKI is its timely recognition. Current diagnostic methods based on serum creatinine, oliguria, or even novel biomarkers, however, take hours to days to become diagnostic. The investigators have no accepted standard for diagnosing kidney hypoxia in real-time before the injury becomes irreversible. Most clinicians base intraoperative hemodynamic goals for the kidney on "educated guesses" of adequate renal perfusion, since the exact cardiac output or mean arterial pressure targets for preventing AKI are unknown. Even the practice of monitoring urine output is uncertain because of its non-specific relationship to kidney function.18-20 Near infrared spectroscopy (NIRS) is a promising technology for monitoring tissue hypoxia because it is noninvasive and has a long history of clinical use as a monitor of cerebral oximetry in both cardiac and vascular surgery. Because NIRS measures a mixture of arterial and venous capillary oxygenation, it is particularly well-suited to monitor the balance between oxygen consumption and delivery. A large body of literature describes the use of NIRS both as a systemic perfusion monitor and a regional monitor of kidney perfusion in neonates and small children.21-26 In adult cardiac surgery patients, two studies using ultrasound guided placement of NIRS sensors over the kidney found that intraoperative regional tissue oxygen desaturations were associated with the subsequent development of AKI.27, 28 A third study found a correlation between NIRS oxygen saturation measurements over the kidney and renal venous oxygen saturation in adult cardiac surgery patients.29 The problem with these studies, however, is that they excluded patients for body mass index (BMI) greater than 30kg/m2 or if the surface of their kidney was greater than 4cm from the skin. According to the Center for Disease Control, the incidence of obesity (BMI greater than 30kg/m2) is over 40% in the United States and obese patients having cardiac surgery are at increased risk for AKI.30, 31 Thus, if NIRS placed over the kidney in adult patients is to be an effective tool in monitoring kidney hypoxia in adults in the United States, then the technology must be effective in all adult patients.

The major limitation to the use of NIRS for renal hypoxia monitoring in adults is the depth of penetration of the signal. Manufacturers guidelines suggest that the maximum depth of penetration of NIRS is 2.5 cm. The actual depth of penetration of NIRS measurements depends on the source-detector separation, the specific algorithm used, and the optical properties of the tissue being measured. When NIRS is modeled experimentally, there is a nonlinear relationship between source-detector separation and depth of penetration such that a source-detector separation of 20 mm resulted in a depth of penetration of 10 mm but a source-detector separation of 40mm resulted in a depth of penetration of 15mm.32 While in very thin adults, the surface of the kidney may be within 2 cm from the skin, the renal medulla (where most AKI is thought to occur) is several centimeters deeper and thus unlikely to be monitored accurately.

The question then arises as to how these adult cardiac surgery studies showed a relationship between NIRS placed over the kidney, AKI outcome, and even renal venous oxygen saturation.27-29 The lab developed a porcine model in which the investigators directly compared kidney medullary oxygen concentration to NIRS measurements placed over the kidney and the thigh during hemorrhagic shock and aortic occlusion.33 The investigators found during extreme hemodynamic changes such as aortic occlusion, there was a moderate correlation between NIRS and invasive kidney tissue oxygen concentration, but this was true irrespective of whether the NIRS sensors were placed over the kidney or over the thigh. The relationship between kidney NIRS and thigh NIRS was stronger than that with kidney oxygen concentration. This was in animals with kidney surface to skin distances of less than 2 cm. Taken together, these data suggest that renal NIRS in adults may be measuring subcutaneous tissue oxygenation but that it is still a global perfusion monitor that may predict poor global perfusion and AKI risk. Indeed, a study in adult cardiac surgery patients showed that NIRS sensors placed over the thigh predicted subsequent AKI with receiver operator characteristic analysis suggesting an optimal cut-off of 67% and an area under the curve of 0.84.34 The purpose of the current study proposal is to directly compare NIRS placed over the kidney to NIRS placed over the arm or the thigh in adult patients having cardiac surgery at risk for AKI. The hypothesis is that limb NIRS and kidney NIRS will both predict AKI and that the ability of NIRS to predict AKI in adult cardiac surgery patients will be independent of BMI and kidney surface to skin distance.

ELIGIBILITY:
Inclusion Criteria:

* We will enroll a convenience sample of adult cardiac surgery patients undergoing procedures that require cardiopulmonary bypass (CPB) and who are at risk for AKI.

Exclusion Criteria:

* Exclusion criteria will include less than age 18 years old, preoperative end-stage kidney disease requiring dialysis, emergency surgery, or patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cardiac surgery patients undergoing procedures that require cardiopulmonary bypass (CPB) and who are at risk for AKI (determined by the Cleveland Risk Score greater than 6) at the University of Utah medical hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Development of post-operative acute kidney injury (AKI) in adult cardiac surgery patients | From post-operative day 0 to post-operative day 7(KDIGO stage I AKI)
  The objective of this study is to compare perioperative renal NIRS and limb NIRS and determine whether these measurements can predict acute kidney injury in adult cardiac surgery patients. The primary outcome will be the as defined by the Kidney Disease: Improving Global Outcomes (KDIGO) guidelines. Measured by an increase in serum creatinine greater than 0.3mg/dl (48 hours) or an increase in serum creatinine greater than 1.5 times baseline (7 days).

SECONDARY OUTCOMES:
The development of severe acute kidney injury (AKI) | From post-operative day 0 to post-operative day 7(KDIGO stage I AKI)
  Post-operative AKI as defined by the Kidney Disease: Improving Global Outcomes (KDIGO) guidelines. Measured by an increase in serum creatinine greater than 2.0 - 2.9 times baseline (KDIGO stage 2) or an increase in serum creatinine greater than 3.0 times baseline or greater than 4mg/dl or the initiation of renal replacement therapy (KDIGO stage 3)
Ventilator times | From post-operative day 0 to end of hospital stay, up to 3 months
  Length of time patient is on ventilator
ICU and hospital length of stay | From post-operative day 0 to end of hospital stay, up to 3 months
  Time patient is in pre-operation (pre-cardiopulmonary bypass(CPB)), operation (CPB), Post-operation (post-CPB), and ICU.
In-hospital mortality | From post-operative day 0 to end of hospital stay, up to 3 months
  Number of in-hospital, operative and/or post-operative (cardiopulmonary bypass) deaths
Intraoperative hemodynamic changes, mean arterial pressure | From start of surgery to end of surgery, up to 24 hours
  Blood pressure (mmHg) readings will be recorded.
Intraoperative hemodynamic changes, oxygen delivery | From start of surgery to end of surgery, up to 24 hours
  Oxygen delivery readings during cardiopulmonary bypass will be recorded (Sp02 using pulse oximeter, measured in liters per minute (LPM)).
Intraoperative hemodynamic changes, vasopressor administration | From start of surgery to end of surgery, up to 24 hours
  Vasopressor agent (mcg/kg/min) use will be recorded.
Intraoperative hemodynamic changes, anemia | From start of surgery to end of surgery, up to 24 hours
  Intraoperative anemia will be measured on both NIRS measurements, expressed as a % (regional SO2 (rS02)).

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Silverton, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No